CLINICAL TRIAL: NCT00798031
Title: Case Series Evaluation of a Short Dental Implant Placed in the Posterior Maxilla in an Early Loading Protocol
Brief Title: Case Series Evaluation of a Short Dental Implant
Acronym: Short implant
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: As of 2017 study was terminated since investigators retired. No subjects recruited.
Sponsor: Clark Stanford (Other)
Responsible Party: Sponsor-Investigator, Clark Stanford, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 200807715
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Tooth Loss
Keywords: dental implant; upper jaw; posterior tooth loss; short dental implant; Adults, 18 years of age and older; Missing a minimum of two posterior teeth in their upper jaw; Subjects in need of dental implants; the research study is survival and function of the implants
MeSH Terms: conditions — Tooth Loss | interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): a minimum of two dental implants, but up to 3 dental implants, will be placed in each of 20 subjects. All surgical procedures will be performed as outpatient procedures at the College of Dentistry and implant placement will follow a one-stage procedure under local anesthesia. Placement of the 2-3 dental implants is the only intervention.
  Interventions: Device: A minimum of two but up to three Astra Tech Dental Implant, Fixture Osseospeed will be placed in the posterior upper jaw of 20 eligible subjects.; Device: Placement of dental implant; Device: dental implant

INTERVENTIONS:
Device: A minimum of two but up to three Astra Tech Dental Implant, Fixture Osseospeed will be placed in the posterior upper jaw of 20 eligible subjects. — A minimum of 2 but up to three dental implants will be placed in the posterior upper jaw of 20 subjects. The dental implants are produced by Astra Tech AB (Fixture Micro Thread OsseoSpeed TM Astra Tech AB. The study will include 15 clinic visits and interim analysis will occur at 6 months, 1, 2, and 3 years after loading of the temporary prosthesis.
  Other Names: Astra Tech AB OsseoSpeed 4mm diameter - 6mm length dental implant; FDA510(k)number: K063779
Device: Placement of dental implant — Device: A minimum of two but up to three Astra Tech Dental Implant, Fixture Osseospeed will be placed in the posterior upper jaw of 20 eligible subjects.
  A minimum of 2 but up to three dental implants will be placed in the posterior upper jaw of 20 subjects. The dental implants are produced by Astra Tech AB (Fixture Micro Thread OsseoSpeed TM Astra Tech AB. the study will include 15 clinic visits and interim analysis will occur at 6 months, 1, 2, and 3 years after loading of the temporary prothesis.
  Other Names: Astra Tech Dental Implant Fixture Osseospeed.; Dental implants are 4.00 mmdiameter x 6mm in length
Device: dental implant — Subjects will have a complete diagnostic work-up performed and assessment for eligibility in the study by both a Prosthodontist and Surgeon. Subjects will then have two and up to three dental implants placed in an out patient basis at the University of Iowa College of Dentistry
  Other Names: 4.0mm diameter x 6 mm in length implant; (Astra Tech Dental Implant, Fixture OsseospeedTM)

SUMMARY:
Following the loss of teeth, the alveolar bone formed in response to the eruption of the teeth is gradually resorbed by the body. In conventional dental implant therapy, a wide safety margin of uninterrupted healing (3-6 months) following placement of the implants is used to assure a predictable survival of the implants (on the order of > 90%). In the past few years, there have been multiple studies documenting with improved implant surface technologies available, that dental implants can be put into function far sooner than conventionally thought. The investigators are currently performing recalls on subjects treated in a research protocol at the University of Iowa (YAOSS-0001; IRB 200305001). Since this initial study, a shortened version of the implant device has been developed and has obtained FDA clearance (FDA 510k 063779 clearance letter dated April 27, 2007) for a 4mm diameter by 6mm in length dental implant. In a case study the investigators are proposing to repeat the same protocol as used in the initial trial with the following exceptions: only this one implant type will be used, no bone compression surgical techniques will be used (referred to as "osteotome" indirect sinus lifting). Our initial trial has documented good performance with minimal bone loss and a 98.3% cumulative survival rate.

This will be an open, prospective case-series clinical documentation study to document the clinical efficacy of the 4.0mm diameter x 6 mm in length implant (Astra Tech Dental Implant, Fixture OsseospeedTM ) in the treatment of subjects missing teeth in the upper jaw. A minimum of two but preferably three implants shall be considered for each surgical site. A total of 20 subjects fulfilling all inclusion criteria will be enrolled. Subjects will have a complete diagnostic work-up performed and assessment for eligibility in the study by both a Prosthodontist and Surgeon. Subjects will then have the implants placed in an out patient basis at the College of Dentistry. The subjects will not wear a conventional removable partial during the initial six weeks of healing. At six weeks, an assessment of the implants shall be made by the surgical and restorative team and if a set of safety benchmarks are met, provisional crowns will be made to place the implants into clinical function (mastication). Over the first year, the provisional crowns will be periodically removed and a series of clinical measurements and mobility measurements made. At the end of 1 year following placement, the permanent crowns or bridgework will be constructed and the subject followed annually for another four years (five years total from placement). A total of 15 clinical visits are estimated per subject.

DETAILED DESCRIPTION:
Subjects will have costs for being in this research study. The costs are for the charges for the dental surgeon who performs the dental implant surgery. Subjects will have a choice of either a College of Dentistry faculty or resident to perform the surgery. The residents are dentists who are receiving specialized training in either Oral Surgery or Periodontics.

If a subject chooses a College of Dentistry Faculty Dentist, the costs are as follows:

For two implants = $4,650.00 For three implants = $6,600.00

If you choose a College of Dentistry Resident Dentist, the costs are as follows:

For two implants = $3,860.00 For three implants = $5,435.00

The dental implant, abutment and false tooth will be provided to each subject at no cost by Astra Tech AB.

If a subject has dental insurance the cost of the surgeon may be covered by your insurance. Potential subjects should check with their insurance carrier regarding coverage prior to agreeing to participate in the research study. Any insurance co-payments that are required will be a cost to the subject.

Methods and Materials This will be an open, prospective case-series clinical documentation study to document the clinical efficacy of the 4.0mm diameter x 6 mm in length implant (Astra Tech Dental Implant, Fixture OsseospeedTM ) in the treatment of subjects missing teeth in the posterior maxilla (referred to as a Kennedy class I or class II situation). A minimum of two but preferably three implants shall be considered for each surgical site. A total of 20 subjects fulfilling all inclusion criteria and none of the exclusions criteria will be enrolled. Bilateral posterior maxilla treatment can be provided (2-3 implants pre-side) but each side must follow the inclusion/exclusion criteria.

The study will be a five-year follow up study with 15 clinic visits. Interim analyses will be performed at 6 months and at 1 and 3 years after loading of the temporary prosthesis.

The study comprises the following three periods:

Pre-surgical evaluation and planning (0 weeks to implant surgery) Surgical and prosthetic treatment (Surgery to 52 weeks/12 months) Follow-up (12 months to 60 months)

The screening procedure will include a clinical and radiographic assessment. Pre-existing radiographs (e.g. panoramic and intraoral periapical images) can be used but must not be older than 6 months. A minimum of 5 mm height (alveolar ridge to sinus floor) is required. Diagnostic steps will involve the fabrication of a surgical guide or surgical denture to indicate the optimal position of the implants for placement in the posterior upper jaw based on the available bone. Preliminary diagnostic impressions will made (Penta, 3M ESPE) and poured in dental stone (Whip Mix Corp., Louisville, KY). Implant subjects may have a pre-operative Cone Bean CT imaging study made at the College of Dentistry's Department of Oral Maxillofacial Radiology at the discretion of the Principal Investigator following diagnostic work-up. Subjects shall be either patients of record of the College of Dentistry or shall be enrolled if new to the College. Patient records will be electronic along with a paper version. Paper-based Case Report Forms (CRF) containing subject's medical information will be kept in one central file in a locked cabinet in the Dental Clinical Research Center. This data will be kept in a secured file accessible only by the PI and the Clinical Coordinator.

Surgical and prosthetic treatment (Surgery to 52 weeks/12 months) Surgical Intervention: All surgical procedures will be performed as outpatient procedures at the College of Dentistry in the Department of Oral and Maxillofacial Surgery or in the Department of Periodontics. Implant placement will follow a one-stage procedure and will be performed under local anesthesia. Prophylactic antibiotic treatment will be given. One hour prior to surgery patients will receive the first dose of a 7 - 10 day prophylactic antibiotic treatment regimen based on Amoxicillin (500mg TID for 7 days) or if allergic to Amoxicillin, Clindamycin (300 mg QID for 7 days). Details of the treatment will be recorded in the clinical case report form (CRF).

Other medication, considered necessary for the patient's welfare, may be given at the discretion of the investigator(s). The administration of all such medication will be recorded in the patient's notes as per normal practice. In addition, medication that may have a negative effect on bone tissue as well as medication to treat any Adverse Event that is considered to be probably or possibly treatment-related must also be recorded in the appropriate sections of the Case Report Form (CRF).

Intravenous conscious sedation is allowed. Conscious out-patient sedation will be "titrated to effect" for the following medications. The dosages will be varied depending upon the subject's age, weight and medical status. Versed (1 to 10 mg.) or Valium (1 to 20 mg.), titrated over the duration of the procedure Fentanyl (0.025 to 0.1 mg) or Demerol (25 to 100 mg), titrated over the duration of the procedure. Phenergan (5 to 25 mg) may be added to either of the narcotics to potentate their effect and extend working time. At the discretion of the surgeon, oral sedation can be used as an alternative (e.g., Valium 5-20mg).

Following achievement of sedation, infiltration of local dental anesthetic is performed [2% Lidocaine HCL with 1:100,000 epinephrine or 4% Atricaine with Epi 1:100,000] immediately prior to surgery. Alternatively, a longer acting local anesthetic [0.5% bupivicaine + 1:200,000 epinephrine] may be used.

In general, all subjects will be treatment planned for a minimum of two implants spaced 7 mm apart (center-to-center) in anatomic regions which will provide sufficient alveolar width for a minimum of 1 mm of bone in all dimensions (minimum of 6 mm ridge width). The objective is to place two to three implants in the upper posterior jaw. Implants will be positioned typically in the anterior residual ridge (below the nasal floor of the maxillary sinus where there is 5 mm or greater than cortical and trabecular bone) and occasionally in the distal wall of the maxillary sinus. Extensive autogenous bone grafting and/or sinus lift grafting will not be performed in this trial. In cases of bilateral edentulism a minimum of two implants will be placed in both locations.

Besides optimal bone support, providing primary stability, the direction/inclination of the implants in the mesiodistal and buccolingual dimensions shall be governed by the requirements for a satisfactory final prosthetic function and esthetics.

Lack of Primary Stability: If an implant does not achieve primary stability, a two stage delayed loading period of 3 months will be performed for all implants placed in this subject.

Use of an osteotome: Localized internal sinus floor elevation with simultaneous implant placement using osteotome technique is not allowed in this protocol.

Cases of sinus perforation will be subjected to standard care of treatment per the investigators discretion and treatment details subsequently recorded in the Case Report From. The surgeon should aim for full bone coverage of the implant threads. Where threads are exposed, augmentation with autogenous bone alone or in combination with Bio-Gide Bilayer Membrane can be used.

Immediately after implant placement (IP) and abutment connection intraoral radiographs of the fixtures will be made and primary stability assessed clinically and by Resonance Frequency Analysis using the OsstellTM device.

The Osstell device is an FDA approved hand held resonance frequency transducer that measures the relative bone stiffness around dental implants. The device consists of a transducer that is connected to the implant or implant abutment and the transducer then applies a small harmonic steady state swept waveform and a second transducer then detects the stiffness of the implant and surrounding bone. The basis of the transducer is an off set cantilever beam (principal of a tuning fork) and the first flexural resonance is then measured. The value of the response is then computed and presented on a scale of 1-100 Implant Stability Quotient (ISQ) value.

Implants will be subjected to a 6-week healing period left in a transmucosal position with the peri-implant mucosa sutured and closely adapted to the abutments. Subjects will not wear a pre-existing removable partial denture over the implant sites during the initial 6 week healing period.

Assessments of implant stability will be evaluated at 6 weeks following placement (Temporary Restoration stage or "TR"), TR +4, 8,12, 26 and 52 weeks respectively.

In cases where primary implant stability cannot be achieved the patient will be treated with a conventional two-stage approach (i.e. submerged healing in combination with an extended healing period of 3 months before uncovering and loading of the implants). Such patient will not be excluded from the study but followed for the full course of the study. During the healing period, patients will be recalled at 2, 4 and 6 weeks following placement. To avoid overloading of the implants, the patient will not be allowed to wear a removable prosthesis over the implants during this period.

TREATMENT OF FAILING IMPLANTS If an implant is lost (fails), as defined below, the site shall be treated in the manner best suited to the well being of the subject. Following implant removal and treatment of the site, the implant may be replaced with another implant or the site may be allowed to heal for future placement of another implant or the site may be allowed to heal without implant replacement. No replacement implants shall be entered into this study. Any implant that is showing excessive bone loss (grater than 5mm), such as radiolucency or infection, shall be treated in the manner best suited to the well-being of the patient, including treatment to save the implant. Treatment may include surgical intervention to resolve infection and/or sequestra and may include administration of topical or systemic antibiotics. Such events and treatments shall be recorded on the Adverse Event form. Implants that are successfully treated shall not be considered treatment failures in this study.

Follow-up (12 months to 60 months) The patient will return for follow-up visits at TR +24, 36, 48 and 60 months. At all follow-up visits evaluation of soft tissue status and treatment related complications will be performed together with intraoral radiographs of the implants.

Radiographic assessments/measurements Intraoral periapical radiographs of the implants will be taken immediately after implant placement, at impression for temporary restoration, at visit 7, visit 8 and visit 9 (12, 26 respectively 52 weeks after implant placement) and at follow-up visits after 24, 36, 48 and 60 months.

The following variables will be recorded:

* periimplant radiolucency will be recorded as presence or absence of radiolucency.
* marginal bone level will be recorded as the vertical distance from the reference point to the marginal bone level. The distance will be measured to the nearest 1/10 mm.

PRIMARY OUTCOMES MEASURES The primary outcome measure in this case series evaluation shall be implant loss (removal).

SECONDARY OUTCOME MEASURE Mobility: A free-standing implant is immobile when tested with instrument pressure. Mobility shall not be quantified. Instead, mobility detectable under the application of pressure by two opposing instruments to an implant shall be considered an indication of failure.

Stability: Implant resonance frequency analysis as measured on the "Implant Stability Quotient" (or ISQ) on a scale of 1-100 will be recorded.

Radiolucency: A standard conventional dental radiograph does not show evidence of continuous peri-implant radiolucency.

Pain, Infection: A successfully integrated implant is characterized by an absence of persistent or irreversible signs and symptoms such as pain and infection.

Bone height: Vertical bone loss of less than 0.2mm annually following the first year of loading.

Patient Adaptation: Patients are satisfied with the esthetics, phonetics and the function of the implant supported crown.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* 18 years of age and over
* Edentulous in the posterior maxilla, Kennedy classes I or II. Last natural tooth, or previously restored implant in function is canine or first premolar.
* Deemed by the investigator as likely to present an initially stabile implant situation suitable for early loading

Exclusion Criteria:

* Untreated caries and/or periodontal disease of residual dentition
* History of edentulism in the area of implant placement of less than two months
* Current need for pre-surgical bone or soft tissue augmentation in the planned implant area.
* History of pre-surgical bone or soft tissue augmentation, within 2 months, in the planned implant area.
* Alveolar bone height of < than 5 mm from the alveolar crest to the floor of the maxillary sinus, verified by periapical radiographs.
* Any systemic or local disease or condition that would compromise post-operative healing and/or osseointegration
* Need for systemic corticosteroids or any other medication that would compromise post-operative healing and/or osseointegration
* Present alcohol or drug abuse
* Unable or unwilling to return for follow-up visits for a period of 5 years
* Current use of smoking tobacco Subjects who require routine antibiotic use for SBE
* Pregnancy or lactation at the time of enrollment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is implant loss (failure). | 6 months and 1, 2 and 3 years after implant loading of the temporary prosthesis

SECONDARY OUTCOMES:
Secondary outcome measure include: mobility, implant stability, peri-implant radiolucency, signs/symptoms of pain or infection, radiographically measured bone loss and patient adaptation. | 6 months, 1, 2, and 3 years after implant loading

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa College of Dentistry, Iowa City, Iowa, United States